CLINICAL TRIAL: NCT02728752
Title: Prospective, Double-blind, Randomized, Placebo-Controlled Phase III Study Evaluating Efficacy and Safety of Octagam 10% in Patients With Dermatomyositis ("ProDERM Study")
Brief Title: Study Evaluating Efficacy and Safety of Octagam 10% in Patients With Dermatomyositis (Idiopathic Inflammatory Myopathy)
Acronym: IIM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GAM10-08
Record Dates: First submitted 2016-03-11; First posted 2016-04-05 (Estimated); Results first posted 2021-04-21 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-11

CONDITIONS: Dermatomyositis
Keywords: DM
MeSH Terms: conditions — Dermatomyositis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects randomized to placebo will receive 4 infusions of placebo every 4 weeks during the blinded First Period (16 weeks). If confirmed deterioration (deterioration at 2 consecutive visits) during the First Period, subjects will be switched to Octagam 10%. After response assessment at Week 16, all subjects with no confirmed deterioration and subjects switched to Octagam 10% due to confirmed deterioration but without further confirmed deterioration during the First Period will continue to receive 2.0 g/kg of Octagam 10% every 4 weeks during the subsequent 6-months open-label Extension Period. At Week 28, subjects who are stable on 2.0 g/kg Octagam 10% can be switched to 1.0 g/kg Octagam 10%, at the discretion of the investigator. Subjects randomized to placebo and switched to Octagam 10% due to confirmed deterioration, who deteriorate also during Octagam 10% treatment at 2 consecutive visits will drop-out after response assessment at Week 16 and will not enter the Extension Period.
  Interventions: Other: Placebo
- Octagam10% (Experimental): Subjects randomized to Octagam will receive 4 infusions of 2.0 g/kg Octagam 10% every 4 weeks during the blinded First Period (16 weeks). If confirmed deterioration (deterioration at 2 consecutive visits) during the First Period, subjects will be switched to the alternate treatment. After response assessment at Week 16, all subjects with no confirmed deterioration during the First Period will continue receiving 2.0 g/kg of Octagam 10% every 4 weeks during the subsequent 6-months open-label Extension Period. At Week 28, subjects who are stable on 2.0 g/kg Octagam 10% can be switched to 1.0 g/kg Octagam 10%, at the discretion of the investigator. Subjects randomized to Octagam and switched to the alternate treatment due to confirmed deterioration will drop-out after response assessment at Week 16 and will not enter the Extension Period.
  Interventions: Drug: Octagam 10%

INTERVENTIONS:
Drug: Octagam 10% — Patients to be treated with Octagam 10%
  Arms: Octagam10%
Other: Placebo — Patients to be treated with a Placebo
  Arms: Placebo

SUMMARY:
Prospective, Double-blind, Randomized, Placebo-Controlled Phase III Study Evaluating Efficacy and Safety of Octagam 10% in Patients With Dermatomyositis ("ProDERM study")

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with diagnosis of definite or probable DM according to the Bohan and Peter criteria.
2. Subjects under treatment with corticosteroids and/or maximally 2 immune-suppressants and being on stable therapy for at least 4 weeks (see Section 4.2.1) OR Subjects with previous failure of response or previous intolerance to corticosteroid and at least 1 additional immunosuppressive drug, and with steroid/immunosuppressive drugs washed out as per Section 4.2.1 (Table 2).
3. Subjects with active disease, assessed and agreed upon by an independent adjudication committee.
4. Manual Muscle Testing-8 (MMT-8) score <142, with at least 2 other abnormal Core Set Measures (CSM) (Visual Analogue Scale [VAS] of patient global activity ≥2 cm, physician's global disease activity ≥2 cm, extra-muscular activity ≥2 cm; at least one muscle enzyme >1.5 times upper limit of normal, Health Assessment Questionnaire ≥0.25).
5. Males or females ≥ 18 to < 80 years of age.
6. Voluntarily given, fully informed written consent obtained from subject before any study-related procedures are conducted.
7. Subject must be capable to understand and comply with the relevant aspects of the study protocol.

Exclusion Criteria:

1. Cancer-associated myositis, defined as the diagnosis of myositis within 2 years of the diagnosis of cancer (except basal or squamous cell skin cancer or carcinoma in situ of the cervix that has been excised and cured and at least 1 or 5 years, respectively, have passed since excision).
2. Evidence of active malignant disease or malignancies diagnosed within the previous 5 years (including hematological malignancies and solid tumors) or breast cancer diagnosed within the previous 10 years.
3. Subjects with overlap myositis (except for overlap with Sjögren's syndrome), connective tissue disease associated DM, inclusion body myositis, polymyositis, juvenile dermatomyositis or drug-induced myopathy.
4. Subjects with immune-mediated necrotizing myopathy with absence of typical DM rash.
5. Subjects with generalized, severe musculoskeletal conditions other than DM that prevent a sufficient assessment of the subject by the physician.
6. Subjects who have received IgG treatment within the last 6 months before enrolment.
7. Subjects who received blood or plasma-derived products (other than IgG) or plasma exchange within the last 3 months before enrolment.
8. Subjects starting or planning to start a physical therapy-directed exercise regimen during the trial.
9. Cardiac insufficiency (New York Heart Association III/IV), cardiomyopathy, significant cardiac dysrhythmia requiring treatment, unstable or advanced ischemic heart disease.
10. Severe liver disease, with signs of ascites and hepatic encephalopathy.
11. Severe kidney disease (as defined by estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2).
12. Known hepatitis B, hepatitis C or HIV infection.
13. Subjects with a history of TEE such as deep vein thrombosis, pulmonary embolism, myocardial infarction, ischemic stroke, transient ischemic attack, peripheral artery disease (Fontaine IV) ever.
14. Body mass index ≥40 kg/m2.
15. Medical conditions whose symptoms and effects could alter protein catabolism and/or IgG utilization (e.g. protein-losing enteropathies, nephrotic syndrome).
16. Known IgA deficiency with antibodies to IgA.
17. History of hypersensitivity, anaphylaxis or severe systemic response to immuno-globulin, blood or plasma derived products or any component of Octagam 10%.
18. Known blood hyperviscosity, or other hypercoagulable states.
19. Subjects with a history of drug abuse within the past 5 years prior to study enrollment.
20. Subjects unable or unwilling to understand or comply with the study protocol.
21. Participating in another interventional clinical study with investigational treatment within 3 months prior to study enrollment.
22. Women who are breast feeding, pregnant, or planning to become pregnant, or are unwilling to apply an effective birth control method (such as implants, injectables, combined oral contraceptives, some intrauterine devices [IUDs], sexual abstinence or vasectomized partner) up to four weeks after the last IMP infusion.
23. Subjects who are accommodated in an institution or care facility based on an official directive or court order.
24. Subjects who are in any way dependent on the Sponsor, Investigator or Study Site.
25. Subjects who received forbidden medication within the washout period as defined in Section 4.2.2 (Table 3).

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Frenzel, Study Director — International Medical Director
Locations (37):
- United States (17):
  - Octapharma Research Site, Huntington Beach, California
  - Octapharma Research Site, Los Angeles, California
  - University of California -Irvine, Orange, California
  - Octapharma Research Site, Orlando, Florida
  - NeuroMedical Research Center, Panama City, Florida
  - Octapharma Research Site, Plantation, Florida
  - University of South Florida, Tampa, Florida
  - Octapharma Research Site, Kansas City, Kansas
  - Octapharma Research Site, Ann Arbor, Michigan
  - Octapharma Research Site, Rochester, Minnesota
  - Octapharma Research Site, Great Neck, New York
  - Octapharma Research Site, Portland, Oregon
  - Octapharma Research Site, Pittsburgh, Pennsylvania
  - Stones River Dermatology, Murfreesboro, Tennessee
  - Austin Neuromuscular Center, Austin, Texas
  - Octapharma Research Site, Houston, Texas
  - Arthritis & Osteoporosis Clinic, Waco, Texas
- Octapharma Research Site, Montreal, Quebec, Canada
- Revmatologický ústav, Prague, Czechia
- Germany (2):
  - Charité-Universitätsmedizin Berlin, Klinik für Dermatologie, Venerologie und Allergologie, Berlin
  - Uniklinikum Münster, Klinik für Hautkrankheiten, Münster
- Hungary (3):
  - Semmelweis University Dermatology Clinic, Budapest
  - University of Debrecen Dept of Internal Medicine, Debrecen
  - University of Szeged Dermatology Clinic, Szeged
- Academic Medical Centre University of Amsterdam, Amsterdam, Netherlands
- Poland (2):
  - Centrum Medyczne Plejady, Krakow
  - Narodowy Instytut Geriatrii, Reumatologii I Rehabilitacji - Warsaw, Warsaw
- Octapharma Research Site, Cluj-Napoca, Romania
- Russia (5):
  - Scientific Research Institute for Rheumatology (Moscow), Moscow
  - I.M. Sechenov First Moscow State Medical University, Moscow
  - Orenburg State Medical University Based On Regional Clinical Hospital, Orenburg
  - 3rd Rheumatology Department Of Clinical Rheumatology Hospital No. 25, Saint Petersburg
  - AVA-Peter clinic (Saint-Petersburg), Saint Petersburg
- Ukraine (4):
  - Octapharma Research Site, Ivano-Frankivsk
  - Octapharma Research Site, Lviv
  - Octapharma Research Site, Sumy
  - Octapharma Research Site, Ternopil

REFERENCES:
- [Derived] Aggarwal R, Schessl J, Bata-Csorgo Z, Dimachkie MM, Griger Z, Moiseev S, Oddis CV, Schiopu E, Vencovsky J, Clodi E, Levine T, Charles-Schoeman C; ProDERM investigators. Efficacy of Intravenous Immunoglobulin for Systemic Manifestations of Dermatomyositis Beyond Muscular and Cutaneous: Sub-analysis of the ProDERM Study. Rheumatol Ther. 2025 Oct;12(5):855-871. doi: 10.1007/s40744-025-00775-5. Epub 2025 Jul 5. PMID 40616720
- [Derived] Charles-Schoeman C, Schessl J, Bata-Csorgo Z, Dimachkie MM, Griger Z, Moiseev S, Oddis CV, Schiopu E, Vencovsky J, Clodi E, Levine T, Aggarwal R. Predictors of response to intravenous immunoglobulin in patients with dermatomyositis: the ProDERM study. Rheumatology (Oxford). 2025 Jun 1;64(6):3767-3776. doi: 10.1093/rheumatology/keaf070. PMID 39918968
- [Derived] Aggarwal R, Schessl J, Charles-Schoeman C, Bata-Csorgo Z, Dimachkie MM, Griger Z, Moiseev S, Oddis CV, Schiopu E, Vencovsky J, Beckmann I, Clodi E, Levine T; ProDERM investigators. Safety and tolerability of intravenous immunoglobulin in patients with active dermatomyositis: results from the randomised, placebo-controlled ProDERM study. Arthritis Res Ther. 2024 Jan 17;26(1):27. doi: 10.1186/s13075-023-03232-2. PMID 38233885
- [Derived] Werth VP, Aggarwal R, Charles-Schoeman C, Schessl J, Levine T, Kopasz N, Worm M, Bata-Csorgo Z. Efficacy of intravenous immunoglobulins (IVIg) in improving skin symptoms in patients with dermatomyositis: a post-hoc analysis of the ProDERM study. EClinicalMedicine. 2023 Oct 2;64:102234. doi: 10.1016/j.eclinm.2023.102234. eCollection 2023 Oct. PMID 37799613
- [Derived] Aggarwal R, Charles-Schoeman C, Schessl J, Bata-Csorgo Z, Dimachkie MM, Griger Z, Moiseev S, Oddis C, Schiopu E, Vencovsky J, Beckmann I, Clodi E, Bugrova O, Danko K, Ernste F, Goyal NA, Heuer M, Hudson M, Hussain YM, Karam C, Magnolo N, Nelson R, Pozur N, Prystupa L, Sardy M, Valenzuela G, van der Kooi AJ, Vu T, Worm M, Levine T; ProDERM Trial Group. Trial of Intravenous Immune Globulin in Dermatomyositis. N Engl J Med. 2022 Oct 6;387(14):1264-1278. doi: 10.1056/NEJMoa2117912. PMID 36198179
- [Derived] Aggarwal R, Charles-Schoeman C, Schessl J, Dimachkie MM, Beckmann I, Levine T. Prospective, double-blind, randomized, placebo-controlled phase III study evaluating efficacy and safety of octagam 10% in patients with dermatomyositis ("ProDERM Study"). Medicine (Baltimore). 2021 Jan 8;100(1):e23677. doi: 10.1097/MD.0000000000023677. PMID 33429735

RESULTS

PARTICIPANT FLOW:
Period: First Period
Arm/Group | Placebo | Octagam10%
Started | 48 | 47
Completed | 46 | 45
Not Completed | 2 | 2
Period: Extension Period
Arm/Group | Placebo | Octagam10%
Started | 46 | 45
Completed | 35 | 34
Not Completed | 11 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Octagam10% | Total
Number analyzed (Participants) | 48 | 47 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.35 (12.979) | 54.04 (13.838) | 52.68 (13.407)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 36 | 71
  Male | 13 | 11 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 43 | 44 | 87
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Measure the Number of Patients Who Had an Increase of ≥20 Points on the Total Improvement Score (TIS)
Description: Proportion of responders in the 2.0 g/kg Octagam 10% and placebo arms at Week 16 relative to baseline (Week 0). A responder being defined as a patient with an increase of ≥20 points on the Total Improvement Score (TIS, a scale from 0 to 100; 20-39 points being minimal improvement, 40-59 points being moderate improvement, and ≥60 points being major improvement
Time Frame: At week 16
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Octagam10%
Number analyzed (Participants) | 48 | 47
Participants | 21 | 37

2. Secondary Outcome: Proportion of TIS Responders by Improvement Category at Week 16
Description: The TIS (Total Improvement Score) is a scale from 0 to 100 that allows for the discrimination between minimal, moderate and major responders depending on their improvement in the combined 6 CSM: ≥20 to 39 points being minimal improvement, ≥40 to 59 points being moderate improvement, and ≥60 points being major improvement.
  Primary: Total number of all patients who had at least minimal, moderate, or major response.
  At Least Moderate: Number of patients who had moderate or major response. At Least Major: Number of patients who had a major response.
Time Frame: 16 weeks
Population: Only responders are displayed as the intent of the outcome measure is to present the proportion of responders. And patients not accounted for were non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Octagam10%
Number analyzed (Participants) | 48 | 47
Participants
  Primary | 21 | 37
  At least moderate improvement | 11 | 32
  At least major improvement | 4 | 15

3. Secondary Outcome: Proportion of TIS Responders by Improvement Category at Week 40
Description: The TIS (Total Improvement Score) is a scale from 0 to 100 that allows for the discrimination between minimal, moderate and major responders depending on their improvement in the combined 6 CSM: ≥20 to 39 points being minimal improvement, ≥40 to 59 points being moderate improvement, and ≥60 points being major improvement.
  At Least Minimal: Total number of all patients who had minimal, moderate, or major response.
  At Least Moderate: Number of patients who had moderate or major response. At Least Major: Number of patients who had a major response.
Time Frame: 40 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Octagam10%
Number analyzed (Participants) | 46 | 45
Participants
  At least minimal improvement | 32 | 32
  At least moderate improvement | 28 | 26
  At least major improvement | 14 | 17

4. Secondary Outcome: Mean Change From Baseline (Week 0) to End of First Period (Week 16) in the Modified Cutaneous Dermatomyositis Disease Area and Severity Index (CDASI)
Description: The modified CDASI has 3 activity measures (erythema, scale, and erosion/ulceration) and 2 damage measures (poikiloderma and calcinosis) which are assessed over 15 body areas. In addition, Gottron's papules on the hands are evaluated both for activity and damage. Lastly, the activity of periungual changes and alopecia is assessed.
  Absence of skin lesions as described above is scored with "0" for each of the above described areas. Skin lesion will be scored with at least "1" (present), some lesions will be graded from "1" (less severe) to "2" (severe); others with "1", "2" or "3". For the total activity score as well as for the total damage score the sub-scores will be added up. The score for total activity ranges from 0 to 100, for total damage from 0 to 32 points. Higher scores indicate greater disease activity or greater disease damage respectively.
Time Frame: First 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Octagam10%
Number analyzed (Participants) | 43 | 45
units on a scale
  Total Activity Score | -1.16 (7.000) | -9.36 (10.542)
  Total Damage Score | -0.02 (0.771) | -0.67 (1.871)
Statistical Analysis 1: Comparison: Placebo vs Octagam10%; LS Means difference between changes from baseline to week 16 for Total Activity Score; Test type: Superiority; p < 0.0001, ANCOVA; With treatment, stratum and baseline as fixed effects, and site as random effect; Mean Difference (Net) = -8.00, 95% CI 2-sided [-11.5 to -4.6] — Difference in LS Means of changes from baseline to week 16 (Octagam - Placebo)

5. Secondary Outcome: Mean Change From End of First Period (Week 16) to End of Extension Period (Week 40) in the Modified Cutaneous Dermatomyositis Disease Area and Severity Index (CDASI)
Description: The modified CDASI has 3 activity measures (erythema, scale, and erosion/ulceration) and 2 damage measures (poikiloderma and calcinosis) which are assessed over 15 body areas. In addition, Gottron's papules on the hands are evaluated both for activity and damage. Lastly, the activity of periungual changes and alopecia is assessed
  Absence of skin lesions as described above is scored with "0" for each of the above described areas. Skin lesion will be scored with at least "1" (present), some lesions will be graded from "1" (less severe) to "2" (severe); others with "1", "2" or "3". For the total activity score as well as for the total damage score the sub-scores will be added up. The score for total activity ranges from 0 to 100, for total damage from 0 to 32 points. Higher scores indicate greater disease activity or greater disease damage respectively.
Time Frame: From week 16 to Week 40
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Octagam10%
Number analyzed (Participants) | 33 | 34
units on a scale
  Total Activity Score | -8.52 (11.344) | -1.79 (4.169)
  Total Damage Score | -0.24 (0.969) | 0.26 (2.220)

6. Secondary Outcome: Mean Change From Baseline (Week 0) to End of Extension Period (Week 40) in the Modified Cutaneous Dermatomyositis Disease Area and Severity Index (CDASI)
Description: as for outcome 4
Time Frame: 40 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Octagam10%
Number analyzed (Participants) | 35 | 34
units on a scale
  Total Activity Score | -10.44 (10.034) | -10.03 (8.995)
  Total Damage Score | -0.26 (1.197) | -0.38 (2.523)

7. Secondary Outcome: Mean Change From Baseline (Week 0) to End of First Period (Week 16) and Extension Period (Week 40) in: SF-36v2 Health Survey
Description: The SF-36 is a multi-purpose, short-form health survey with only 36 questions. It yields an 8-scale profile of functional health and well-being scores as well as psychometrically-based physical and mental health summary measures and a preference-based health utility index.
  SF-36 scores ranging from 0 to 100. 0 represented the lowest possible score (worst health state) and 100 represented the highest possible score (best health state), with scores in between representing the percentages of the total possible score achieved by respondents on a given scale.
Time Frame: From start of the trial till Week 40
Population: Numbers of patients analyzed different due to patient discontinuations through study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Octagam10%
Number analyzed (Participants) | 43 | 43
units on a scale
  Baseline to Week 16 | 2.27 (4.598) | 7.06 (8.220)
  Baseline to Week 40: number analyzed (Participants) | 35 | 34
  Baseline to Week 40 | 6.65 (8.258) | 8.77 (10.930)

8. Secondary Outcome: Mean Change From Baseline (Week 0) to End of First Period (Week 16) and Extension Period (Week 40) in Physician's Global Disease Activity
Description: 10 cm VAS assessing global disease activity from "No evidence of disease activity" to "Extremely active or severe disease activity"; Disease Activity being defined as potentially reversible pathology or physiology resulting from the myositis). Assessment completed by physician. 0 is lowest score and 10 is highest score. Higher score associated with worse outcome.
Time Frame: From start of the trial till Week 40
Population: Different numbers of patients analyzed in each group due to patient discontinuation.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Octagam10%
Number analyzed (Participants) | 43 | 45
score on a scale
  Baseline to Week 16 | -0.60 (1.815) | -2.39 (1.987)
  Baseline to Week 40: number analyzed (Participants) | 35 | 34
  Baseline to Week 40 | -2.93 (1.888) | -3.06 (1.817)

9. Secondary Outcome: Mean Change From Baseline (Week 0) to End of First Period (Week 16) and Extension Period (Week 40) in: Patient Global Disease Activity
Description: Patient's Global Disease Activity (10cm VAS assessing the overall activity of the patient's disease today from "No evidence of disease activity" to "Extremely active or severe disease activity", Disease Activity being active inflammation in the patient's muscles, skin, joints, intestines, heart, lungs or other parts of the body, which can improve when treated with medicines). 0 is lowest score and 10 is highest score. Higher score associated with worse outcome.
Time Frame: From start of the trial till Week 40
Population: Different numbers of patients analyzed in each group due to patient discontinuation.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Octagam10%
Number analyzed (Participants) | 43 | 45
score on a scale
  Baseline to Week 16 | -1.11 (2.094) | -2.19 (2.276)
  Baseline to Week 40: number analyzed (Participants) | 35 | 33
  Baseline to Week 40 | -2.77 (2.133) | -2.71 (2.651)

10. Secondary Outcome: Mean Change From Baseline (Week 0) to End of First Period (Week 16) and Extension Period (Week 40) in: MMT-8
Description: Manual Muscle Testing - MMT-8; a set of 8 designated muscles tested bilaterally [potential score 0 - 150]. Higher score associated with better outcome.
Time Frame: From start of the trial till Week 40
Population: Different numbers of patients analyzed in each group due to patient discontinuation.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Octagam10%
Number analyzed (Participants) | 43 | 45
score on a scale
  Baseline to Week 16 | 3.21 (9.390) | 14.38 (14.581)
  Baseline to Week 40: number analyzed (Participants) | 35 | 33
  Baseline to Week 40 | 12.00 (7.491) | 20.09 (14.486)
Statistical Analysis 1: Comparison: Placebo vs Octagam10%; LS Means difference between changes from baseline to week 16; Test type: Superiority; p = 0.0001, ANCOVA; With treatment, stratum and baseline as fixed effects, and site as random effect; Median Difference (Net) = 8.6, 95% CI 2-sided [4.4 to 12.8] — Difference in LS Means of changes from baseline to week 16 (Octagam - Placebo)

11. Secondary Outcome: Mean Change From Baseline (Week 0) to End of First Period (Week 16) and Extension Period (Week 40) in: Health Assessment Questionnaire
Description: Health Assessment Questionnaire (HAQ); a generic rather than a disease-specific instrument; comprised of 8 sections: dressing, arising, eating, walking, hygiene, reach, grip, and activities. There are 2 or 3 questions for each section. Scoring within each section is from 0 [without any difficulty] to 3 [unable to do]. For each section the score given to that section is the worst score within the section. The 8 scores of the 8 sections are summed and divided by 8). Assessment completed by patients. Lowest score 0 highest score 24. Higher score associated with worse outcome.
Time Frame: From start of the trial till Week 40
Population: Different numbers of patients analyzed in each group due to patient discontinuation.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Octagam10%
Number analyzed (Participants) | 43 | 45
score on a scale
  Baseline to Week 16 | -0.16 (0.366) | -0.56 (0.590)
  Baseline to Week 40: number analyzed (Participants) | 34 | 33
  Baseline to Week 40 | -0.54 (0.524) | -0.66 (0.805)
Statistical Analysis 1: Comparison: Placebo vs Octagam10%; LS Means difference between changes from baseline to week 16; Test type: Superiority; p = 0.0002, ANCOVA; With treatment, stratum and baseline as fixed effects, and site as random effect; Median Difference (Net) = -0.4, 95% CI 2-sided [-0.5 to -0.2] — Difference in LS Means of changes from baseline to week 16 (Octagam - Placebo)

12. Secondary Outcome: Mean Change From Baseline (Week 0) to End of First Period (Week 16) and Extension Period (Week 40) in Enzymes (Alanine Aminotransferase)
Time Frame: From start of the trial till Week 40
Population: Different numbers of patients analyzed in each group due to patient discontinuation.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | Octagam10%
Number analyzed (Participants) | 43 | 42
U/L
  Baseline to Week 16 | -4.47 (29.796) | -8.52 (18.474)
  Baseline to Week 40: number analyzed (Participants) | 35 | 33
  Baseline to Week 40 | -4.06 (14.787) | -7.15 (18.480)

13. Secondary Outcome: Mean Change From Baseline (Week 0) to End of First Period (Week 16) and Extension Period (Week 40) in Enzymes (Aspartate Aminotransferase)
Time Frame: From start of the trial till Week 40
Population: Different numbers of patients analyzed in each group due to patient discontinuation.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | Octagam10%
Number analyzed (Participants) | 43 | 44
U/L
  Baseline to Week 16 | -3.07 (31.317) | -7.82 (26.139)
  Baseline to Week 40: number analyzed (Participants) | 35 | 34
  Baseline to Week 40 | -2.20 (16.421) | -7.76 (26.431)

14. Secondary Outcome: Mean Change From Baseline (Week 0) to End of First Period (Week 16) and Extension Period (Week 40) in Enzymes (Lactate Dehydrogenase)
Time Frame: From start of the trial till Week 40
Population: Different numbers of patients analyzed in each group due to patient discontinuation.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | Octagam10%
Number analyzed (Participants) | 43 | 45
U/L
  Baseline to Week 16 | -19.79 (142.012) | -11.04 (165.252)
  Baseline to Week 40: number analyzed (Participants) | 35 | 34
  Baseline to Week 40 | -33.43 (63.651) | -59.21 (92.801)

15. Secondary Outcome: Mean Change From Baseline (Week 0) to End of First Period (Week 16) and Extension Period (Week 40) in Enzymes (Aldolase)
Time Frame: From start of the trial till Week 40
Population: Different numbers of patients analyzed in each group due to patient discontinuation.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | Octagam10%
Number analyzed (Participants) | 41 | 42
U/L
  Baseline to Week 16 | -2.51 (12.077) | -0.48 (7.743)
  Baseline to Week 40: number analyzed (Participants) | 35 | 32
  Baseline to Week 40 | -0.59 (7.839) | -1.48 (3.644)

16. Secondary Outcome: Mean Change From Baseline (Week 0) to End of First Period (Week 16) and Extension Period (Week 40) in Enzymes (Creatine Kinase)
Time Frame: From start of the trial till Week 40
Population: Different numbers of patients analyzed in each group due to patient discontinuation.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | Octagam10%
Number analyzed (Participants) | 43 | 44
U/L
  Baseline to Week 16 | -352.79 (2141.534) | -169.20 (434.224)
  Baseline to Week 40: number analyzed (Participants) | 35 | 34
  Baseline to Week 40 | -56.54 (556.928) | -169.38 (449.210)

17. Secondary Outcome: Mean Change From Baseline (Week 0) to End of First Period (Week 16) and Extension Period (Week 40) in: Extra-muscular Activity
Description: 10 cm VAS assessing extra-muscular activity from "No evidence of disease activity" to "Extremely active or severe disease activity". It encompasses an overall evaluation for the disease activity in all the extramuscular organ systems and excludes muscle disease activity. Assessment completed by physician. 0 is lowest score and 10 is highest score. Higher score associated with worse outcome.
Time Frame: From start of the trial until Week 40
Population: Different numbers of patients analyzed in each group due to patient discontinuation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Octagam10%
Number analyzed (Participants) | 43 | 45
units on a scale
  Baseline to Week 16 | -0.94 (2.287) | -2.18 (2.134)
  Baseline to Week 40: number analyzed (Participants) | 35 | 34
  Baseline to Week 40 | -2.64 (2.092) | -2.67 (2.061)
Statistical Analysis 1: Comparison: Placebo vs Octagam10%; LS Means difference between changes from baseline to week 16; Test type: Superiority; p = 0.0010, ANCOVA; With treatment, stratum and baseline as fixed effects, and site as random effect; Median Difference (Net) = -1.2, 95% CI 2-sided [-1.9 to -0.5] — Difference in LS Means of changes from baseline to week 16 (Octagam - Placebo)

18. Secondary Outcome: Mean TIS From Baseline (Week 0) to End of First Period (Week 16) and From Baseline (Week 0) to End of Extension Period (Week 40)
Description: The TIS (Total Improvement Score) is a scale from 0 to 100 that allows for the discrimination between minimal, moderate and major responders depending on their improvement in the combined 6 CSM: ≥20 to 39 points being minimal improvement, ≥40 to 59 points being moderate improvement, and ≥60 points being major improvement.
Time Frame: Up to 40 weeks
Population: Different numbers of patients analyzed in each group due to patient discontinuation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Octagam10%
Number analyzed (Participants) | 43 | 45
units on a scale
  Week 16 | 21.57 (20.185) | 48.44 (24.444)
  Week 40: number analyzed (Participants) | 35 | 34
  Week 40 | 51.07 (18.314) | 55.44 (21.712)

19. Secondary Outcome: Time to Minimal, Moderate and Major Improvement in TIS
Description: When interpreting these time to event evaluations, one has to keep in mind that eventually all patients were treated with octagam 10%, so that differences in time to response for the Overall Period reflect this delayed start of treatment rather than the true difference between treatment with octagam 10% and placebo.
Time Frame: Up to 40 weeks
Population: Number of participants based on number of responders. 95% confidence interval not available for all measurements.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Octagam10%
Number analyzed (Participants) | 48 | 47
days
  Time to Minimal Improvement - First Period: number analyzed (Participants) | 23 | 42
  Time to Minimal Improvement - First Period | 115.0 [84.0 to NA] — Insufficient number of participants with events | 35.0 [29.0 to 58.0]
  Time to Moderate Improvement - First Period: number analyzed (Participants) | 11 | 34
  Time to Moderate Improvement - First Period | NA [NA to NA] — Insufficient number of participants with events | 85.0 [58.0 to 113.0]
  Time to Major Improvement - First Period: number analyzed (Participants) | 5 | 15
  Time to Major Improvement - First Period | NA [NA to NA] — Insufficient number of participants with events | NA [115.0 to NA] — Insufficient number of participants with events
  Time to Minimal Improvement - From Start of First Treatment in Overall Period: number analyzed (Participants) | 41 | 47
  Time to Minimal Improvement - From Start of First Treatment in Overall Period | 114.0 [84.0 to 195.0] | 35.0 [29.0 to 58.0]
  Time to Moderate Improvement - From Start of First Treatment in Overall Period: number analyzed (Participants) | 36 | 39
  Time to Moderate Improvement - From Start of First Treatment in Overall Period | 197.0 [195.0 to 282.0] | 85.0 [58.0 to 113.0]
  Time to Major Improvement - From Start of First Treatment in Overall Period: number analyzed (Participants) | 20 | 25
  Time to Major Improvement - From Start of First Treatment in Overall Period | 283.0 [203.0 to NA] — Insufficient number of participants with events | 283.0 [197.0 to 290.0]

20. Secondary Outcome: Time to Confirmed Deterioration in the First Period and Overall
Description: Confirmed deterioration is defined as disease worsening on 2 consecutive visits. Worsening criteria are defined as either Physician's Global Disease Activity worsening ≥2cm and Manual Muscle Testing worsening ≥20% or Extra-muscular Activity worsening ≥2cm or any 3 of the following scores worsening by ≥30%: Physician's Global Disease Activity, Manual Muscle Test, Extra-muscular Activity, Patient's Global Disease Activity or Health Assessment Questionnaire.
Time Frame: Up to 40 weeks
Population: All patients analyzed and only those that had confirmed deterioration are presented.
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Octagam10%
Number analyzed (Participants) | 3 | 1
days
  First Period: number analyzed (Participants) | 3 | 0
  First Period | 58 [57 to 117] |
  Overall Period | 58 [57 to 117] | 142 [NA to NA] — Single participant

ADVERSE EVENTS:
Time Frame: 40 weeks
Description: Note that the AE tables summarize data by the actual treatment at the time of the AE. An AE was considered to be associated with the most recent treatment administered, octagam 10% or placebo. Patients who were switched to the alternate treatment during the First Period were therefore considered to be 'at risk' for AEs in both treatment groups.
Groups:
- First Period Placebo: Subjects randomized to placebo will receive 4 infusions of placebo every 4 weeks during the blinded First Period (16 weeks). If confirmed deterioration (deterioration at 2 consecutive visits) during the First Period, subjects will be switched to Octagam 10%. After response assessment at Week 16, all subjects with no confirmed deterioration and subjects switched to Octagam 10% due to confirmed deterioration but with not further confirmed deterioration during the First Period will continue to receive 2.0 g/kg of Octagam 10% every 4 weeks during the subsequent 6-months open-label Extension Period. At Week 28, subjects who are stable on 2.0 g/kg Octagam 10% can be switched to 1.0 g/kg Octagam 10%, at the discretion of the investigator. Subjects randomized to placebo and switched to Octagam 10% due to confirmed deterioration, who deteriorate also during Octagam 10% treatment at 2 consecutive visits will drop-out after response assessment at Week 16 and will not enter the Extension Period.
- Overall Period Octagam: Subjects randomized to Octagam will receive 4 infusions of 2.0 g/kg Octagam 10% every 4 weeks during the blinded First Period (16 weeks). If confirmed deterioration (deterioration at 2 consecutive visits) during the First Period, subjects will be switched to the alternate treatment. After response assessment at Week 16, all subjects with no confirmed deterioration during the First Period will continue receiving 2.0 g/kg of Octagam 10% every 4 weeks during the subsequent 6-months open-label Extension Period. At Week 28, subjects who are stable on 2.0 g/kg Octagam 10% can be switched to 1.0 g/kg Octagam 10%, at the discretion of the investigator. Subjects randomized to Octagam and switched to the alternate treatment due to confirmed deterioration will drop-out after response assessment at Week 16 and will not enter the Extension Period.
Arm/Group | First Period Placebo | Overall Period Octagam
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/95
Serious Adverse Events (participants affected / at risk) | 2/48 | 14/95
Other Adverse Events (participants affected / at risk) | 28/48 | 84/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | First Period Placebo (N=48) | Overall Period Octagam (N=95)
Sinus tachycardia (Cardiac disorders) | 1 (2) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Tropical spastic paresis (Infections and infestations) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Condition aggravated (General disorders) | 0 (0) | 2 (2)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | First Period Placebo (N=48) | Overall Period Octagam (N=95)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 2 (2) | 1 (2)
Mitral valve calcification (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2) | 5 (6)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Pulmonary valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 4 (7)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 18 (30)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 9 (12)
Asthenia (General disorders) | 1 (1) | 3 (7)
Catheter site erythema (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 2 (2)
Chest pain (General disorders) | 3 (3) | 3 (3)
Chills (General disorders) | 1 (2) | 7 (12)
Condition aggravated (General disorders) | 9 (22) | 9 (13)
Extravastation (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 4 (4) | 5 (6)
Feeling cold (General disorders) | 1 (1) | 0 (0)
Infusion site bruising (General disorders) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 2 (4)
Malaise (General disorders) | 0 (0) | 1 (2)
Oedema peripheral (General disorders) | 0 (0) | 3 (3)
Pain (General disorders) | 0 (0) | 2 (3)
Peripheral swelling (General disorders) | 1 (1) | 3 (3)
Pyrexia (General disorders) | 3 (3) | 17 (26)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Asymptomatic bacteriuria (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 3 (3)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 6 (8)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 3 (4)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 2 (2) | 0 (0)
Blood potassium increased (Investigations) | 1 (1) | 0 (0)
Blood pressure decreased (Investigations) | 0 (0) | 1 (1)
Blood pressure diastolic increased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 3 (4) | 4 (8)
Blood pressure systolic increased (Investigations) | 0 (0) | 3 (3)
Blood urea increased (Investigations) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 5 (8)
Coombs test positive (Investigations) | 0 (0) | 5 (5)
Haemoglobin decreased (Investigations) | 1 (1) | 4 (5)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 7 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (6)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 9 (12)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basilar artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 5 (6)
Headache (Nervous system disorders) | 4 (10) | 46 (102)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urine abnormality (Renal and urinary disorders) | 0 (0) | 1 (7)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Diffuse alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (6)
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Essential hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 5 (6)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Peripheral coldness (Vascular disorders) | 0 (0) | 1 (2)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Eye disorder (Eye disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1)
Infusion site pain (General disorders) | 0 (0) | 1 (1)
Infusion site reaction (General disorders) | 0 (0) | 1 (1)
Infusion site swelling (General disorders) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 0 (0) | 1 (1)
Injection site induration (General disorders) | 0 (0) | 1 (1)
Local swelling (General disorders) | 0 (0) | 1 (2)
Nodule (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 2 (3)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Lyme disease (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (3)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2)
Cardiac murmur (Investigations) | 0 (0) | 1 (1)
Free haemoglobin present (Investigations) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 0 (0) | 1 (1)
Muscle enzyme increased (Investigations) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (9)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Poikiloderma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Urticaria contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Menopause (Social circumstances) | 0 (0) | 1 (1)
Postmenopause (Social circumstances) | 0 (0) | 1 (1)
Brachiocephalic arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Infusion site erythema (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/52/NCT02728752/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/52/NCT02728752/SAP_001.pdf